Desoximetasone 0.25% Shampoo

Protocol / Study No. DSXS 1536 / 71515013

### STATISTICAL ANALYSIS PLAN

A Randomized, Double-Blind, Vehicle-Controlled, Parallel-Design, Multiple-Site, Phase III Clinical Study to Evaluate the Efficacy and Safety of Desoximetasone 0.25% Shampoo in Patients with Mild to Severe Scalp Psoriasis

Protocol Number: DSXS 1536 Novum Study Number: 71515013

### **Sponsor:**

Taro Pharmaceuticals U.S.A., Inc. 3 Skyline Drive, Hawthorne, NY 10532 USA

### **Contract Research Organization:**

Novum Pharmaceutical Research Services 225 W. Station Square Drive, Suite 200 Pittsburgh, PA 15219

October 11, 2016

Final Version 1.0

Desoximetasone 0.25% Shampoo

Protocol / Study No. DSXS 1536 / 71515013

### SAP FINAL VERSION APPROVALS

A Randomized, Double-Blind, Vehicle-Controlled, Parallel-Design, Multiple-Site, Phase III Clinical Study to Evaluate the Efficacy and Safety of Desoximetasone 0.25% Shampoo in Patients with Mild to Severe Scalp Psoriasis

| Written By: Signature: Jianhua Liu, MSc Senior Biostatistician Novum Pharmaceutical Research Services | Date: 10/13/2016 |
|---|---|
| Reviewed By: Signature: Pina D'Angelo, MSc Senior Director, Scientific Affairs (Biostatistics) Novum Pharmaceutical Research Services | Date: Oct 13, 2016 |
| Approved By: Signature: NYantorskiy Natalie Yantovskiy Senior Director, Clinical Research Taro Pharmaceuticals U.S.A., Inc. | Date: 12 October 2016 |

Desoximetasone 0.25% Shampoo Protocol / Study No. DSXS 1536 / 71515013

# **Revision History**

| Version | DATE | DESCRIPTION OF REVISIONS | REVISED BY |
|---|---|---|---|
| Draft 1.0 | October 03, 2016 | New Document | Jianhua Liu |
| Final 1.0 | October 11, 2016 | Incorporate client comments and finalize SAP | Jianhua Liu |

### Desoximetasone 0.25% Shampoo

Protocol / Study No. DSXS 1536 / 71515013

### List of Abbreviations and Definition of Terms

ADaM Analysis Data Model

AE Adverse Event BP Blood Pressure

C Celsius

CRF Case Report Form

CDISC Clinical Data Interchange Standards Consortium

CRO Contract Research Organization

F Fahrenheit

FDA Food and Drug Administration HEENT Head, Eyes, Ears, Nose, Throat

Hg Mercury

ICF Informed Consent Form

ICH International Conference on Harmonization

IGA Investigator's Global Assessment

IND Investigational New Drug

LOCF Last Observation Carried Forward

MedDRA Medical Dictionary for Regulatory Activities

ITT Intent-to-Treat

OGD The Office of Generic Drugs
SAE Serious Adverse Event
SAP Statistical Analysis Plan
SAS Statistical Analysis System
SDTM Study Data Tabulation Model
USA United States of America

# Desoximetasone 0.25% Shampoo Protocol / Study No. DSXS 1536 / 71515013

### TABLE OF CONTENTS

| 1. | INTRODUCTION | 7 |
|---|---|---|
| 2. | OBJECTIVES | 7 |
| 3. | OVERALL STUDY DESIGN | 7 |
| 4. | RANDOMIZATION AND BLINDING | 10 |
| 5. | SAMPLE SIZE | 10 |
| 6. | STUDY ENDPOINTS | 11 |
| 7. | STUDY POPULATIONS | 11 |
| 8. | STATISTICAL ANALYSIS METHODS | 11 |
| | 8.1 Baseline Characteristics | 11 |
| | 8.1.1 Patient Disposition | 11 |
| | 8.1.2 Demographic and Other Baseline Characteristics | 12 |
| | 8.1.3 Medical History | |
| | 8.1.4 Concomitant Medications | |
| | 8.2 Efficacy Analyses | 13 |
| | 8.2.1 Primary Analysis | |
| | 8.2.2 Sensitivity Analyses | |
| | 8.3 Safety Analysis | |
| | 8.3.1 Adverse Events | |
| | 8.3.2 Vital Signs | 14 |
| | 8.3.3 Skin Safety Assessments | 14 |
| | 8.3.4 Ocular Discomfort Assessment | 14 |
| | 8.4 Multiple Comparisons | 15 |
| | 8.5 Methods for Handling Missing Data | 15 |
| | 8.6 Interim Analyses | 15 |
| 9. | TABLE, LISTING AND FIGURE SHELLS | 15 |
| | T16.1.9.1 Summary of Patient Disposition | 17 |
| | T16.1.9.2 Summary of Protocol Deviations | 18 |
| | T16.1.9.3.1 Summary of Patients Excluded from Efficacy Analysis (Population | |
| | Determination) | 19 |
| | T16.1.9.3.2 Summary of Patients Included in Analysis Population by Study Center | |
| | T16.1.9.4 Summary of Demographic Data (Safety Population) | 21 |
| | T16.1.9.5 Summary of Demographic Data (Intent-to-Treat Population) | 22 |
| | T16.1.9.6 Summary of Frequency of Investigator Global Assessment (IGA) (Intent- | |
| | to-Treat Population) | 23 |
| | T16.1.9.7 Summary of Analysis Results of Proportion of Patients in each Treatment | |
| | that Have Clinical Success at Visit 3 (Day 29±2) (Intent-to-Treat Population) | 24 |
| | T16.1.9.8 Sensitivity Testing 1: Summary of Analysis Results of Proportion of | |
| | Patients in each Treatment that Have Clinical Success at Visit 3 (Day 29±2) | |
| | (Intent-to-Treat Population) | 25 |

### Desoximetasone 0.25% Shampoo Protocol / Study No. DSXS 1536 / 71515013

| T16.1.9.9 Sensitivity Testing 2: Summary of Analysis Results of Proportion of | |
|---|---|
| Patients in each Treatment that Have Clinical Success at Visit 3 (Day 29±2) (Intent-to-Treat Population) | 26 |
| T16.1.9.10 Summary of Percent Scalp Affected with Scalp Psoriasis by Visit (Intent- | 20 |
| to-Treat Population)to-Treat Population | 27 |
| T16.1.9.11 Overall Summary of Adverse Events | 28 |
| T16.1.9.12 Summary of Frequency of All Adverse Events by Body System (Safety | |
| | 29 |
| T16.1.9.13 Summary of Frequency of All Adverse Events by Body System with | |
| Frequency $\geq 2\%$ in Any Treatment Group (Safety Population) | 20 |
| T16.1.9.14 Summary of Frequency of All Adverse Events by Relationship (Safety | 2 |
| | 30 |
| T16.1.9.15 Summary of Frequency of All Adverse Events by Severity (Safety | |
| Population) | 31 |
| T16.1.9.16 Summary of Frequency of Serious Adverse Events (Safety Population) | |
| T16.1.9.17 Summary of Vital Signs (Safety Population) | |
| T16.1.9.18 Summary of Skin Irritation Assessment (Safety Population) | |
| L16.2.1 Listing of Discontinued Patients | |
| L16.2.2 Listing of Protocol Deviations | |
| L16.2.3 Patients Excluded from the Analysis Population | 37 |
| L16.2.4.1 Listing of Demographic Data | 38 |
| L16.2.4.2 Listing of Medical History | 39 |
| L16.2.4.3 Listing of Concomitant Medication | 40 |
| L16.2.5.1 Listing of Drug Administration | |
| L16.2.5.2 Listing of Study Medication Weight | |
| L16.2.6.1 Listing of Investigator Global Assessment (IGA) | |
| L16.2.6.2 Listing of Percent Scalp Affected with Scalp Psoriasis | |
| L16.2.7.1 Listing of Adverse Events by Treatment | |
| L16.2.7.2 Listing of Skin Irritation Assessment | |
| L16.2.7.3 Listing of Ocular Signs/Symptoms Assessment | |
| L16.2.7.4 Listing of Positive Pregnancy Test Results | |
| L16.2.7.5 Listing of Abnormal Physical Examinations | |
| 10. APPENDICES | 50 |
| Appendix A: Investigator's Global Assessment (IGA) of Disease Severity of Scalp | |
| Psoriasis | |
| Appendix B: Skin Assessment (Forehead, Neck and Ears) | |
| Appendix C: Ocular Discomfort Assessment | 52 |

Desoximetasone 0.25% Shampoo Protocol / Study No. DSXS 1536 / 71515013

### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) is based on the final Clinical Study Protocol DSXS 1536 (Novum Study No. 71515013) Rev. 2 dated 05/31/2016. The SAP provides details on the planned statistical methodology for the analysis of the study data. The SAP also outlines the statistical programming specifications for the tables, listings and figures.

This SAP describes the study endpoints, derived variables, anticipated data transformations and manipulations, and other details of the analyses not provided in the study protocol. This SAP therefore outlines in detail all other aspects pertaining to the planned analyses and presentations for this study.

The following documents were reviewed in preparation of this SAP:

- Final Clinical Study Protocol DSXS 1536 (Novum Study No. 71515013) Rev. 2 dated 05/31/2016
- Case Report Form Booklet Version 1.0 for Novum Study No. 71515013 dated 03/03/2016

The reader of this SAP is encouraged to also read the clinical protocol for details on the conduct of this study, and the operational aspects of clinical assessments and timing for completing a patient in this study.

### 2. OBJECTIVES

The objective of this study is to evaluate the therapeutic efficacy and safety of desoximetasone 0.25% shampoo (Taro Pharmaceuticals, U.S.A., Inc.) compared to a Vehicle shampoo (Taro Pharmaceuticals, U.S.A., Inc.) in patients with mild to severe scalp psoriasis.

### 3. OVERALL STUDY DESIGN

This randomized, double-blind, vehicle-controlled, parallel-group multiple-site study is designed to evaluate the therapeutic efficacy and safety of the investigational product, desoximetasone 0.25% shampoo (Taro Pharmaceuticals, U.S.A.), for the treatment of mild to severe scalp psoriasis.

Up to 370 eligible patients with scalp psoriasis that satisfy all eligibility criteria will be enrolled into the study at Visit 1. Patients must be at least 18 years of age, in overall good health. They should have a current diagnosis of mild to severe scalp psoriasis with IGA score of at least 2.

Patients who meet all inclusion/exclusion criteria will be randomized in a 1:1 ratio (Test: Vehicle) at Visit 1. At least 185 qualified patients will receive Test product and 185 patients will receive Vehicle product. The product will be left in place on the scalp for 15 minutes.

### Desoximetasone 0.25% Shampoo

Protocol / Study No. DSXS 1536 / 71515013

At Visit 1, patients who meet all inclusion/exclusion criteria will be randomized in a 1:1 ratio (Test: Vehicle) for 28 days of treatment:

The study products are:

- Test: Desoximetasone 0.25% Shampoo (Taro)
- Vehicle: Test Vehicle Shampoo (Taro)

Patients in each randomized treatment group will apply product once daily, according to provided instructions, for a total of 28 days starting on Day 1.

During the study patients will visit the clinical center for a total of 3 scheduled visits:

- Visit 1 (Day -1 to 1): Randomization
- Visit 2 (Day  $14 \pm 2$ ): Interim Visit
- Visit 3 (Day  $29 \pm 2$ ): End of Study or Early Termination

The primary efficacy endpoint is the proportion of patients in each treatment group who are considered a Clinical Success, as defined by an IGA score of 0 (clear) or 1 (almost clear) with at least a 2-grade improvement from baseline IGA at Day  $29 \pm 2$ . That is, at Day  $29 \pm 2$ , patients with an IGA score of 3 or 4 at baseline must achieve a score of 0 or 1, patients with an IGA score of 2 at baseline must achieve a score of 0 to be considered a Clinical Success. The 5-point IGA score represents an overall severity of scalp psoriasis based on plaque elevation, scaling and erythema. Severity represented by a score of 0-4 is categorized as 'clear', 'minimal', 'mild', 'moderate' or 'severe'. Refer to Appendix A for IGA scoring.

The safety profile of each treatment group will be evaluated by comparing adverse events, dermal and ocular discomfort and vital signs obtained through the study duration.

Desoximetasone 0.25% Shampoo Protocol / Study No. DSXS 1536 / 71515013

Figure 1 Study Schematic

| Figure 1 Study Schema | Visit 1 | Visit 2 | Visit 3 |
|---|---|---|---|
| Day | -1 to 1 | 14 ± 2 | 29 ± 2 |
| Procedures | Baseline/Rand omization <sup>†</sup> | Interim<br>Visit | End of Study |
| Informed Consent | X | | |
| Medical History and<br>Baseline Demographics | X | | |
| Inclusion/Exclusion | X | | |
| Physical Examination | X | | X |
| HEENT Examination | X | X | X |
| Vital Signs | X | X | X |
| Pregnancy Test* | X | X | X |
| Percent Scalp Affected | X | X | X |
| Investigator's Global<br>Assessment | X | X | X |
| Skin Assessment | X | X | X |
| Ocular Discomfort<br>Assessment | | X | X |
| Concomitant<br>Medications | X | X | X |
| Weigh and Dispense<br>Study Product | X | X | |
| Collect and Weigh<br>Study Product | | X | X |
| Review/Provide Patient<br>Diary | X | X | X |
| Adverse Events | | X | X |

<sup>\*</sup> Pregnancy test will be conducted for females of childbearing potential.

<sup>†</sup> Patients should administer study product once daily for 28 days starting on Day 1 through Day 28. The product will be left in place on the scalp for 15 minutes.

Desoximetasone 0.25% Shampoo Protocol / Study No. DSXS 1536 / 71515013

### 4. RANDOMIZATION AND BLINDING

At Visit 1 eligible patients will be randomized to the study and assigned a randomization number. Patient numbers will consist of a 2-digit site number and 4-digit randomization number. The 4-digit randomization numbers will be assigned in ascending order beginning with the lowest number at each study site.

The study product will be packaged and blinded by an independent clinical packaging company. The randomization will be generated in blocks of 4 to accommodate the 1:1 randomization scheme (2 Test:2 Vehicle).

Each eligible patient will receive 2 x 120 ml bottles of study product (Test or Vehicle). Patients will be randomized to a treatment group in a blinded fashion by assigning randomization numbers in ascending sequential order starting with the lowest available randomization number at each site. All patients randomized will be identified by initials, date of birth, and a unique sixdigit patient number. A perforated two-part label will be attached to each of the small sized boxes of study product supplies. Both pieces of the label will include the following information: Protocol number, randomization number, dosing instructions, space for patient's initials, statement that the study product is for investigational use only, space for dispensing date and the Sponsor's name. One part of the label shall remain attached to the box. The other part will be removed prior to dispensing and attached to the patient source documents. In addition all patients will be provided with written instructions on how to use the study product. Prior to dispensing, study product will be weighed.

At the end of the study, after all the clinical data has been entered and the study database has been locked, a copy of the randomization will be sent to the statistician.

The Investigator, staff at the study site, study monitors, and data analysis/management personnel will be blinded to the patient assignment.

### 5. SAMPLE SIZE

The primary statistical analysis of interest is a comparison of clinical success, as defined by an IGA score of 0 (clear) or 1 (almost clear) with at least 2 grades reduction from baseline at Day  $29 \pm 2$ , of the Test treatment, desoximetasone 0.25% shampoo, to the clinical success of the respective Vehicle shampoo in the ITT population. Based on results from Taro's Phase II study 71342608, the clinical success of the Test formulation is expected to be approximately 27% for an application duration of 15 minutes. The clinical success of the Vehicle formulation is expected to be approximately 10% for the same application duration. Based on a two-sided, Yates' continuity-corrected Z-test and a pooled response rate for the standard error of the difference in proportions, 166 patients in the active group and 166 patients in the placebo group of the ITT population will provide at least 97% power to demonstrate superiority at the 5% significance level (p < 0.05) for the active treatment over placebo. To allow for about 10% of patients who may drop out from the study or are otherwise non-evaluable, up to 370 patients may be enrolled (185 in the active group and 185 in the placebo group).

### Desoximetasone 0.25% Shampoo

Protocol / Study No. DSXS 1536 / 71515013

### 6. STUDY ENDPOINTS

The primary efficacy endpoint is the proportion of patients in each treatment group who are considered a Clinical Success at Day  $29 \pm 2$ , as defined by an IGA score of 0 (clear) or 1 (almost clear) with at least a 2 grades reduction from baseline at Day  $29 \pm 2$ . That is, at Day  $29 \pm 2$ , patients with an IGA score of 3 or 4 at baseline must achieve a score of 0 or 1 and patients with an IGA score of 2 at baseline must achieve a score of 0 to be considered a Clinical Success.

### 7. STUDY POPULATIONS

### **Intent-to-Treat (ITT) Population**

The ITT population will include:

• All randomized subjects.

### **Safety Population**

• All patients who were randomized and applied at least one dose of the study product.

### 8. STATISTICAL ANALYSIS METHODS

If not otherwise specified, statistical significance is defined as p<0.05 and is two-tailed. Data will be summarized with respect to demographic and baseline characteristics and safety variables.

For categorical variables, the number and percent of each category within a parameter will be calculated for non-missing data. For continuous variables, statistics will include n, mean, standard deviation, median, minimum and maximum values.

All statistical analyses will be conducted using SAS<sup>®</sup>, Version 9.4 or higher. Datasets will be prepared using headings from Clinical Data Interchange Consortium (CDISC) Study Data Tabulation Model (SDTM) implementation for human clinical trials and ADaM (Analysis Dataset Model).

### 8.1 Baseline Characteristics

### 8.1.1 Patient Disposition

The patient disposition information will be summarized by treatment. The number of patients randomized, treated with study medication will be tabulated by treatment. In addition, completion status and primary reason for withdrawal will be summarized by treatment.

### Desoximetasone 0.25% Shampoo

Protocol / Study No. DSXS 1536 / 71515013

### 8.1.2 Demographic and Other Baseline Characteristics

Baseline comparability of all treatment groups will be evaluated separately in the ITT and Safety populations.

The following baseline demographics (determined from their initial study visit) will be evaluated:

- Age (years)
- Gender (male/female)
- Ethnicity (Hispanic/non Hispanic)
- Race (White, Black/African American, Native Hawaiian or Other Pacific Islander, Asian, American Indian or Alaska Native, Other)
- % Scalp affected
- Number of months and/or years patient has suffered from symptoms caused by scalp psoriasis

Summary tables by treatment will be presented. Continuous variables will be summarized using descriptive statistics (n, mean, standard deviation, median, minimum, maximum). Categorical variables will be summarized using frequencies and percentage.

Baseline comparability of the treatments will be presented using Chi-square test for the categorical variables, and Analysis of Variance for the continuous variables.

All data will be listed by treatment and patient.

### 8.1.3 Medical History

At Visit 1, patients will be questioned about personal medical history, including acute and chronic medical history and medical history relevant to their scalp psoriasis, as well as all medication use within the past 24 weeks.

Medical history data will be listed by treatment and patient.

### **8.1.4 Concomitant Medications**

At each clinic visit, patients will be questioned about current and concomitant medication use. Patients will also be questioned about ongoing or new concomitant medication use during the treatment period at Visits 2 and 3.

All prior and concomitant medications taken since screening until the end of the study will be listed by treatment and patient.

### Desoximetasone 0.25% Shampoo

Protocol / Study No. DSXS 1536 / 71515013

### 8.2 Efficacy Analyses

### 8.2.1 Primary Analysis

Superiority of the Test shampoo over the Vehicle shampoo at Day  $29 \pm 2$  will be tested using a two-sided Cochran-Mantel-Haenszel (CMH) test, stratified by clinical site, at the 5% significance level. The primary analysis will be performed using Last Observation Carried Forward (LOCF) approach.

Patients discontinued because of lack of treatment effect will be included in the primary analysis as treatment failures.

### 8.2.2 Sensitivity Analyses

The following two sensitivity analyses will also be performed on the primary efficacy endpoint:

- 1. Primary analysis will be performed also including patients without an assessment at Day  $29 \pm 2$ . Patients with missing data at Day  $29 \pm 2$  will be considered clinical failures.
- 2. Primary analysis will be performed also including patients without an assessment at Day  $29 \pm 2$ . Patients from the Vehicle group with missing data at Day  $29 \pm 2$  will be treated as clinical successes and patients from the Test group with missing data at Day  $29 \pm 2$  will be treated as clinical failures.

### 8.3 Safety Analysis

Safety analysis will be conducted on safety population.

### 8.3.1 Adverse Events

All the adverse events (AEs) reported throughout the study will be coded and classified according to the MedDRA (Medical Dictionary for Regulatory Activities) coding dictionary (Version 18.1 or higher). Each adverse event is to be evaluated for date of start and end, seriousness, severity, causal relationship with the study drugs, action taken and outcome.

All AEs will be listed by treatment and patient.

A summary table of the number and percent of patients with AEs by system organ class, preferred term, and treatment will be presented. Each patient will be counted only once within each preferred term. Other summaries may be added based on the obtained data.

A frequency summary table of the number of AEs by system organ class, preferred term, severity, and treatment will be presented. Severity will be classified as "Mild", "Moderate", or "Severe".

### Desoximetasone 0.25% Shampoo

Protocol / Study No. DSXS 1536 / 71515013

Similarly, a frequency summary table of the number of AEs by system organ class, preferred term, and relationship to a study drug, and treatment will be presented. Relationship to a study drug will be classified as "Not Related" or "Related" where "Related includes "Possible", "Probable", or "Definite".

Should sufficient data exist, adverse event frequencies will be compared between treatments using Fisher's exact test.

### 8.3.2 Vital Signs

The patient's vital signs will be recorded (pulse rate, blood pressure, temperature and respiration rate) at Visit 1, 2 and 3.

Descriptive summaries (number of observations, mean, standard deviation, minimum, median and maximum) will be provided by treatment and visit.

All data will be listed by treatment and patient.

### 8.3.3 Skin Safety Assessments

As a part of safety evaluation at each clinic visit, the Investigator/designated clinician will conduct an careful assessment of the scalp and adjacent skin (e.g., ears, forehead and neck) for local tolerability and a score will be documented (refer to Appendix B).

A summary table of the number and percent of patients with different dermal response score will be presented by visit and treatment group.

All data will be listed by patient and visit.

### 8.3.4 Ocular Discomfort Assessment

Ocular discomfort will be assessed by subjects and reported to clinic staff during scheduled visits (refer to Appendix C). If the shampoo comes into contact with the patient's eyes, the patient will be asked to report the contact at each visit.

Ocular safety evaluations will be assessed at the discretion of the Investigator based on the findings of the HEENT exam performed at each visit along with the ocular discomfort reported by the patient. Medical records associated with the ocular safety evaluation should be obtained for the study chart.

Ocular discomfort assessment will be listed by patient and visit.

Desoximetasone 0.25% Shampoo

Protocol / Study No. DSXS 1536 / 71515013

### 8.4 Multiple Comparisons

No multiple comparison adjustment will be made in this study.

### 8.5 Methods for Handling Missing Data

For demographic and baseline characteristics, each variable will be analyzed using all available data. Patients with missing data will be excluded only from analyses for which data are not available.

The primary analysis will be performed using Last Observation Carried Forward (LOCF) approach.

Patients discontinued because of lack of treatment effect will be included in the primary analysis as treatment failures.

### 8.6 Interim Analyses

There is no interim analysis planned in this study.

### 9. TABLE, LISTING AND FIGURE SHELLS

The following shells are provided in order to provide a framework for the display of data from this study. These shells may not be reflective of every aspect of this study but are intended to show the general layout of the Tables, Listings and Figures that will be included in the final clinical study report. Tables, Listings and Figures are numbered following the ICH structure. Table headers, variables names and footnotes will be modified as needed following data analyses. All descriptive and inferential statistical analyses will be performed using SAS® statistical software Version 9.4 or higher, unless otherwise noted.

TABLE, LISTING AND FIGURE SHELLS


T16.1.9.1 Summary of Patient Disposition

Novum Pharmaceutical Research Services Protocol / Study No. DSXS 1536 / 71515013

| | Test | Vehicle | |
|--------------------------|----------------|--------------|-------|
| Patients | Desoximetasone | Test Vehicle | Total |
| | 0.25% Shampoo | Shampoo | |
| Screened | | | XXX |
| Randomized | xxx | XXX | XXX |
| Completed Study | xxx | XXX | XXX |
| Terminated Early | xxx | XXX | XXX |
| Early Termination Reason | ×× | XXX | XXX |
| Adverse Event | XXX | XXX | XXX |
| Lack of Efficacy | XXX | XXX | XXX |
| Lost to follow-up | XXX | XXX | XXX |
| etc. | | | |
| Other | XXX | XXX | XXX |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm

T16.1.9.2 Summary of Protocol Deviations

Novum Pharmaceutical Research Services Protocol / Study No. DSXS 1536 / 71515013

| | Test Desoximetasone 0.25% Shampoo | Vehicle<br>Test Vehicle Shampoo | Total |
|---|---|---|---|
| Total Patients with Protocol Deviations | XXX | XXX | XXX |
| Total Deviations | XXX | XXX | xxx |
| Dosed more than twice on any particular day | XXX | XXX | XXX |
| Failure to meet randomization criteria | XXX | XXX | XXX |
| Lost to Follow-up | XXX | XXX | XXX |
| Missed Visit | XXX | XXX | XXX |
| Missed 4 or more consecutive doses | XXX | XXX | XXX |
| Non-compliance with study drug | XXX | XXX | XXX |
| Outside Visit Window | XXX | XXX | XXX |
| Restricted Medication Use | XXX | XXX | XXX |
| Other | XXX | XXX | XXX |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm


T16.1.9.3.1 Summary of Patients Excluded from Efficacy Analysis

# (Population Determination)

| | Test<br>Desoximetasone<br>0.25% Shampoo | Vehicle<br>Test Vehicle<br>Shampoo | Total |
|---|---|---|---|
| Randomized / ITT Population | XXX | XXX | xxx |
| Safety Population | XXX | XXX | xxx |
| Excluded from Safety population | xxx | XXX | XXX |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm


Taro Pharmaceuticals U.S.A., Inc Desoximetasone 0.25% Shampoo

T16.1.9.3.2 Summary of Patients Included in Analysis Population by Study Center

Novum Pharmaceutical Research Services Protocol / Study No. DSXS 1536 / 71515013

| | Total | ××× | XXX |
|--------|-----------------------------------------|------|------|
| Safety | Vehicle<br>Test Vehicle<br>Shampoo | XXX | XXX |
| | Test Desoximetasone 0.25% Shampoo | XXX | XXX |
| | Total | XXX | XXX |
| LLL | | XXX | XXX |
| | Test<br>Desoximetasone<br>0.25% Shampoo | XXX | XXX |
| | Total<br>Randomized | XXX | XXX |
| | Name | XXXX | XXXX |
| | Site<br>No. | × | × |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm

T16.1.9.4 Summary of Demographic Data

(Safety Population)

| | | Test Desoximetasone 0.25% Shampoo N=xx | Vehicle<br>Test Vehicle<br>Shampoo<br>N=xx | Total<br>N=xx | P-value |
|---|---|---|---|---|---|
| Age (years) | u | XX | XX | XX | X.XXXX |
| | Mean ± SD | $XX.X \pm X.X$ | $XX.X \pm X.X$ | $XX.X \pm X.X$ | |
| | Median | xx.x | XX.X | xx.x | |
| | Range | XX-XX | XX-XX | XX-XX | |
| Race | American Indian or Alaska Native | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | X.XXXX |
| | Asian | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Black/African American | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Native Hawaiian or other Pacific<br>Islander | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | White | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Ethnicity | Hispanic or Latino | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | X.XXXX |
| | Not Hispanic or Latino | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Gender | Female | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | X.XXXX |
| | Male | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

N= number of patients in the treatment; n= number of patient with data available; % is based on N

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm


T16.1.9.4 Summary of Demographic Data (continued) (Safety Population)

| | | Test Desoximetasone 0.25% Shampoo N=xx | Vehicle<br>Test Vehicle<br>Shampoo<br>N=xx | Total<br>N=xx | P-value |
|---|---|---|---|---|---|
| Percent Scalp Affected | u | XX | XX | XX | X.XXXX |
| | Mean ± SD | $XX.X \pm X.X$ | $XX.X \pm X.X$ | $xx.x \pm x.x$ | |
| | Median | XX.X | XX.X | XX.X | |
| | Range | XX-XX | XX-XX | XX-XX | |
| Number of months and/or years patient has suffered from symptoms caused by scalp psoriasis | S months | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XXXXX |
| | >3 months and <6 months | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | >6 months and ≤1 year | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | >1 year and ≤3 years | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | >3 years and <5 years | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | >5 years | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

N= number of patients in the treatment; n= number of patient with data available; % is based on N

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm


Similar tables will be created for T16.1.9.5

T16.1.9.5 Summary of Demographic Data (Intent-to-Treat Population)

Taro Pharmaceuticals U.S.A., Inc Desoximetasone 0.25% Shampoo

T16.1.9.6 Summary of Frequency of Investigator Global Assessment (IGA) (Intent-to-Treat Population)

| | | Test | Vehicle |
|---------------------------|--------------|----------------|--------------|
| 7:0:4 | 3,00 | Desoximetasone | Test Vehicle |
| VISIL | Score | 0.25% Shampoo | Shampoo |
| | | N=xx | N=xx |
| Visit 1 | 0 (Clear) | xx (xx.x%) | (%x.xx) xx |
| | 1 (Minimal) | xx (xx.x%) | xx (xx.x%) |
| | 2 (Mild) | xx (xx.x%) | xx (xx.x%) |
| | 3 (Moderate) | xx (xx.x%) | xx (xx.x%) |
| | 4 (Severe) | xx (xx.x%) | xx (xx.x%) |
| Visit 2 | 0 (Clear) | XX (XX.X%) | xx (xx.x%) |
| | 1 (Minimal) | xx (xx.x%) | xx (xx.x%) |
| | 2 (Mild) | xx (xx.x%) | xx (xx.x%) |
| | 3 (Moderate) | xx(xx.x%) | xx (xx.x%) |
| | 4 (Severe) | xx (xx.x%) | xx (xx.x%) |
| Visit 3/Early termination | 0 (Clear) | xx (xx.x%) | xx (xx.x%) |
| | 1 (Minimal) | xx (xx.x%) | xx (xx.x%) |
| | 2 (Mild) | xx(xx.x%) | xx (xx.x%) |
| | 3 (Moderate) | xx (xx.x%) | xx (xx.x%) |
| | 4 (Severe) | xx (xx.x%) | xx (xx.x%) |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm


T16.1.9.7 Summary of Analysis Results of Proportion of Patients in each Treatment that Have Clinical Success (Intent-to-Treat Population) at Visit 3 (Day 29±2)

| Treatment | Number of | Number of Patients with | Proportion of Patients with | Test vs | Test vs. Vehicle |
|---|---|---|---|---|---|
| Group | Patients (N) | Clinical Success (n). | Clinical Success (%) | Difference P-value | P-value |
| Vehicle | xxx | XXX | XX.X% | | |
| Test | XXX | XXX | %x.xx | %X.XX | X.XXX |

Superiority of Test over Placebo was tested using a two-sided Cochran-Mantel-Haenszel (CMH) test, stratified by clinical site, at the 5% significance level using last observation carried forward (LOCF).

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm

Protocol / Study No. DSXS 1536 / 71515013

T16.1.9.8 Sensitivity Testing 1: Summary of Analysis Results of Proportion of Patients in each Treatment that Have Clinical Success at Visit 3 (Day 29±2) (Intent-to-Treat Population)

| Treatment | Number of | Number of Patients with | Proportion of Patients with | Test vs | Test vs. Vehicle |
|---|---|---|---|---|---|
| Group | Patients (N) | Clinical Success (n) | Clinical Success (%) | Difference P-value | P-value |
| Vehicle | xxx | XXX | %X.XX | | |
| Test | xxx | XXX | xx.x% | xx.x% | X.XXXX |

Superiority of Test over Placebo was tested using a two-sided Cochran-Mantel-Haenszel (CMH) test, stratified by clinical site, at the 5% significance level. Patients with missing data at Day  $29 \pm 2$  will be considered clinical failures.

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm


T16.1.9.9 Sensitivity Testing 2: Summary of Analysis Results of Proportion of Patients in each Treatment that Have Clinical Success at Visit 3 (Day 29±2)

(Intent-to-Treat Population)

| Treatment | Number of | Number of Number of Patients with | Proportion of Patients with | Test vs | Test vs. Vehicle |
|---|---|---|---|---|---|
| Group | Patients (N) | Clinical Success (n) | Clinical Success (%) | Difference P-value | P-value |
| Vehicle | XXX | XXX | %x.xx | | |
| Test | XXX | XXX | xx.x% | %X.XX | X.XXXX |

Superiority of Test over Placebo was tested using a two-sided Cochran-Mantel-Haenszel (CMH) test, stratified by clinical site, at the 5%

significance level. Patients from the Vehicle group with missing data at Day  $29 \pm 2$  will be treated as clinical successes and patients from the Test group with missing data at Day  $29 \pm 2$  will be treated as clinical failures.

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm


T16.1.9.10 Summary of Percent Scalp Affected with Scalp Psoriasis by Visit

(Intent-to-Treat Population)

| | | Test | Vehicle |
|---------------------------|------------|------------------|------------------|
| 45 - 57 M | Statistic. | Desoximetasone | Test Vehicle |
| VISIT | Statistic | 0.25% Shampoo | Shampoo |
| | | N=xx | N=xx |
| Visit 1 | и | ×× | XX |
| | Mean ± SD | $xxx.x \pm xx.x$ | $XXX.X \pm XX.X$ |
| | Median | XXXX.X | XXX.X |
| | Range | xxx - xxx | XXX - XXX |
| Visit 2 | u | XX | XX |
| | Mean ± SD | $xxx.x \pm xx.x$ | $XXX.X \pm XX.X$ |
| | Median | XXXX.X | XXX.X |
| | Range | xxx - xxx | XXX - XXX |
| Visit 3/Early termination | п | XX | XX |
| | Mean ± SD | $xxx.x \pm xx.x$ | $XXX.X \pm XX.X$ |
| | Median | XXXX.X | XXX.X |
| | Range | XXX - XXX | XXX - XXX |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm

Taro Pharmaceuticals U.S.A., Inc Desoximetasone 0.25% Shampoo

T16.1.9.11 Overall Summary of Adverse Events

| Description | l est<br>Desoximetasone<br>0.25% Shampoo<br>N=xx | Venicle<br>Test Vehicle<br>Shampoo<br>N=xx | Total<br>N=xx |
|---|---|---|---|
| Patients Randomized | XXX | XXX | XXX |
| Patients with at least one AE | xx (xx.x%) | xx (xx.x%) | (0/X.XX) |
| Discontinued study drug due to above AEs | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| AEs reported | XXX | XXX | XXX |
| Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Moderate | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not Related | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Related | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx |
| Death | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Serious AE | (%X:XX) XX | (%x.xx) xx | xx (xx.x%) |

Related = "Possible", "Probable", or "Definite" related.

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm

Protocol / Study No. DSXS

T16.1.9.12 Summary of Frequency of All Adverse Events by Body System (Safety Population)

| | | | Test | Ve | Vehicle | |
|---|---|---|---|---|---|---|
| | | Desoxi | Desoximetasone | Test | Fest Vehicle | |
| | | 0.25% | 0.25% Shampoo | Sha | Shampoo | |
| | | | N=xx | Z | N=xx | |
| Body System | MedDRA Term Events Patients | Events | Patients | Events | Events Patients | Fisher's<br>p-value |
| Patients with at least one AE Total | Total | XX | (%x.xx) xx | XX | (%x.xx) xx | X.XXXX |
| Ear and labyrinth disorders | Ear pain | ×× | xx (xx.x%) | XX | xx (xx.x%) | X.XXXX |
| | etc. | | | | | |
| etc. | | | | | | |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm


Repeat table T16.1.9.12 for frequency  $\geq 2\%$  in any treatment group

T16.1.9.13 Summary of Frequency of All Adverse Events by Body System with Frequency ≥ 2% in Any Treatment Group (Safety Population)


T16.1.9.14 Summary of Frequency of All Adverse Events by Relationship

(Safety Population)

| (Saicty a opulation) | Test Vehicle Desoximetasone Test Vehicle | 0.25% Shampoo Shampoo # of Events | $(\mathbf{x}\mathbf{x}\mathbf{x}) \qquad \qquad (\mathbf{x}\mathbf{x}\mathbf{x})$ | Related Not Related Not Related | (x(x,x,%) x(x,x,%) x(x,x,%) x(x,x,%) x(x,x,%) | xx (xx.x%) $xx (xx.x%)$ $xx (xx.x%)$ $xx (xx.x%)$ | xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) |
|---|---|---|---|---|---|---|---|
| | | | | Body System MedDRA Term | Total | Ear and labyrinth Ear pain x> | Hypoacusis |

N = Total number of events in each treatment group; Percentage is based on total number of events. Related includes "Possible", "Probable", or "Definite" related.

Path: L:\Studies\_Sas\_Codes\Clinical Tria\\71515013\PDF\xxx Created on: ddmmmyy hh:mm

T16.1.9.15 Summary of Frequency of All Adverse Events by Severity (Safety Population)

| Vehicle Test Vehicle Shampoo # of Events (N = xxx) Mild Moderate xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) | Vehicle Test Vehicle Shampoo # of Events (N = xxx) Mild Moderate x (xx.x%) xx (xx.x%) x (xx.x%) xx (xx.x%) x (xx.x%) xx (xx.x%) | | MedDRA Term Total Ear pain | Body System Total AEs Ear and labyrinth disorders |
|---|---|---|---|---|
| xx (xx.x%) xx (xx.x%) xx (xx.x%) | ( (xx.x%) xx (xx. | $X = (\%X.XX) \times (\%X.XX) \times (\%X.XX) \times X$ | Hypoacusis | |
| (%x.xx) xx (%x. | (xx.x%) xx (xx. | | Ear pain | Ear and labyrinth disorders |
| (%x.xx) xx (%x. | xx.x%) xx (xx.xx. | | Total | Total AEs |
| rate Severe | Mild Mode | | MedDRA Term | Body System |
| xxx) | (N) | (N = xxx) | | |
| vents | # of E | # of Events | | |
| 00dι | Shan | 0.25% Shampoo | | |
| ehicle | Test V | Desoximetasone | | |
| icle | Veh | Test | | |
| | | (Saicty robulation) | | |

N = Total number of events in each treatment group; Percentage is based on total number of events.

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm


T16.1.9.16 Summary of Frequency of Serious Adverse Events

(Safety Population)

| | | Test | Vehicle |
|---|---|---|---|
| Doder Suctom | ModDRA Torm | Desoximetasone | l est Vehicle |
| Dody System | | 0.25% Shampoo | Shampoo |
| | | # Events | # Events |
| Injury, poisoning and procedural complications | Alcohol poisoning | XX | XX |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmnyy hh:mm


T16.1.9.17 Summary of Vital Signs

| (Safety Population) | | |
|---------------------|---|------|
| Popu | | |
| Popu | • | 2 |
| | • | Ξ |
| | | 2 |
| (Safe | | |
| S | • | Ę |
| | • | 2101 |

| Vital Signs | Visit | Statistic | Test Desoximetasone 0.25% Shampoo | Vehicle<br>Test Vehicle<br>Shampoo<br>N=xx |
|---|---|---|---|---|
| Systolic Blood Pressure (mmHg) | Visit 1 | u | xx | XX |
| | | Mean ± SD | $xxx.x \pm xx.x$ | $XXX.X \pm XX.X$ |
| | | Median | xxx.x | XXXX.X |
| | | Range | XXX - XXX | XXX - XXX |
| | Visit 2 | | | |
| | Visit 3/Early termination | | | |

Diastolic Blood Pressure (mmHg)
Pulse rate (bpm)

Respiration Rate (rpm) Temperature (F) Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm

■ Taro Pharmaceuticals U.S.A., Inc ■


T16.1.9.18 Summary of Skin Irritation Assessment

Taro Pharmaceuticals U.S.A., Inc Desoximetasone 0.25% Shampoo (Safety Population)

| | | Test | Vehicle |
|---------|----------|----------------|--------------|
| | | Desoximetasone | Test Vehicle |
| | Response | 0.25% Shampoo | Shampoo |
| Visit | Score | N=xx | N=xx |
| Visit 1 | (N) 0 | xxx (xx.x%) | xxx (xx.x%) |
| | (Z) - | xxx (xx.x%) | xxx (xx.x%) |
| | 1 (A) | xxx (xx.x%) | xxx (xx.x%) |
| | etc | xxx (xx.x%) | xxx (xx.x%) |

Visit 3/Early termination Visit 2


Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm

# Taro Pharmaceuticals U.S.A., Inc Desoximetasone 0.25% Shampoo

| Novum Pharmaceutical Research Services | Protocol / Study No. DSXS 1536 / 71515013 |
|---|---|

Test Vehicle Shampoo

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm

L16.2.2 Listing of Protocol Deviations

| T | Patient | | |
|---|---|---|---|
| I rearment | Randomization | Event Description | Population |
| Group | Number | | |
| Desoximetasone 0.25% Shampoo | XXXX-XX | Outside Visit Window (Visit 3) | Safety |

Test Vehicle Shampoo


Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm

■ Taro Pharmaceuticals U.S.A., Inc ■


L16.2.3 Patients Excluded from the Analysis Population

| 1 | Patient | Included in | Reason. If Not | Included in | Reason. If Not |
|---|---|---|---|---|---|
| I reatment | Randomization Safety | n Safety | Included in | ITI | Included in ITT |
| Group | Number | Population? | Safety Population | Population? | Population |
| Desoximetasone 0.25% Shampoo | XXXX-XX | Ves | XXXXXXXXX | No<br>No | XXXXXXXXXX |
| | \\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\ | 3 | | | |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm


■ Taro Pharmaceuticals U.S.A., Inc ■

Taro Pharmaceuticals U.S.A., Inc Desoximetasone 0.25% Shampoo

L16.2.4.1 Listing of Demographic Data

| reatment<br>Group | atient<br>Randomization<br>Number | Age | Gender | Ethnicity | Race |
|---|---|---|---|---|---|
| Desoximetasone 0.25% Shampoo | XXXX-X | 30 | Female | Not Hispanic or Latino | Black or African American |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm


Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm

# L16.2.4.2 Listing of Medical History

| Ongoing | |
|---------------------------------------|---------------------------------|
| End Date | yyyy-mm-dd |
| Start Date | yyyy-mm-dd |
| Diagnosis or<br>Surgical<br>Procedure | Menopause |
| System | Gynecologic |
| Patient<br>Randomization<br>Number | xxxx-xx |
| Treatment<br>Group | Desoximetasone 0.25%<br>Shampoo |

Test Vehicle Shampoo


L16.2.4.3 Listing of Concomitant Medication

Test: Desoximetasone 0.25% Shampoo

| | | 1 | | | | | |
|---|---|---|---|---|---|---|---|
| Patient<br>Randomization<br>Number | Treatment<br>Area | Medication | Dosage | Frequency Route | Route | Start/End<br>Date | Indication |
| XX-XXX | No<br>No | Lisinopril | 20 MG QD | | PO | yyyy-mm-dd /<br>yyyy-mm-dd | Hypertension |

Table will continue for vehicle group.

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm

L16.2.5.1 Listing of Drug Administration

| Treatment | Patient | Date of | Date of | Total | Compliance |
|---|---|---|---|---|---|
| , | Randomization | First Dosa | I act Doce | Doses | (%) |
| Group | Number | THE DOSC | Last Dosc | Applied | (6/) |
| Desoximetasone 0.25% Shampoo | XXXX | pp-mm-xxxx | pp-mm-aaa | × | XX.X |
| | | | , , | | |

Compliance = [Actual number of applications] / [Planned number of applications] \* 100%, where: Programming notes:

Planned number of applications is determined as follows:

for patients who completed the study successfully: 28 applications (28 days of once daily dosing); for patients who discontinued early: the minimum between 28 and (Date of Discontinuation – Date of First Application +1).

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm


L16.2.5.2 Listing of Study Medication Weight

Novum Pharmaceutical Research Services Protocol / Study No. DSXS 1536 / 71515013

| | Patient | Bottle | le 1 | Bottle 2 | le 2 | Total |
|---|---|---|---|---|---|---|
| I reatment<br>Group | Randomization<br>Number | Weight<br>Dispensed | Weight<br>Collected | Weight<br>Dispensed | Weight<br>Collected | Dose<br>Used |
| | | (g) | (g) | (g) | (g) | (g) |
| Desoximetasone 0.25% Shampoo | XXXX | XX | X | XX | XX | XX |

Test Vehicle Shampoo

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm

### Taro Pharmaceuticals U.S.A., Inc Desoximetasone 0.25% Shampoo

L16.2.6.1 Listing of Investigator Global Assessment (IGA)

Novum Pharmaceutical Research Services Protocol / Study No. DSXS 1536 / 71515013

| Treatment Patient Randomizatio Group Number | zation | Visit 1 | Visit 2 | Visit 3 / Early<br>Termination | Clinical<br>Success |
|---|---|---|---|---|---|
| Desoximetasone 0.25% Shampoo xx-xxxx | | Mild | Mild | Clear | Yes |
| XXXX-XX | | Clear | Mild | Mild | No |

Test Vehicle Shampoo

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm

L16.2.6.2 Listing of Percent Scalp Affected with Scalp Psoriasis

| | D | • | 1 | |
|---|---|---|---|---|
| Treatment<br>Group | Patient<br>Randomization<br>Number | Visit | Percent Scalp Affected with Scalp Psoriasis | Number of Months or Years<br>the Patient has Suffered from<br>Symptoms of Scalp Psoriasis |
| Desoximetasone 0.25% Shampoo | xxxx | Visit 1 | %xxx | X.XX |
| | • | Visit 2<br>Visit 3/Early Termination | %xxx | |


Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013 \PDF\xxx Created on: ddmmmyy hh:mm


L16.2.7.1 Listing of Adverse Events by Treatment

| | | Test: De | Test: Desoximetasone 0.25% Shampoo | 0.25% Sh | 1ampoo | | | |
|---|---|---|---|---|---|---|---|---|
| atient<br>Randomization<br>Vumber | Body System /<br>MedDRA Term /<br>AE Term | Treatment Start/End<br>Area Date | Start /End<br>Date | Severity | Relationship<br>Severity to Study<br>Drug | Outcome Action<br>Taken | | Other<br>Action<br>Taken |
| (X-XXX | Nervous system disorders / No | / No | yyyy-mm-dd / Mild | Mild | Possible | Recovered Dose Not None | e Not | Vone |
| | Headache / | | yyyy-mm-dd | | | Cha | Changed | |
| | Headache | | | | | | | |

SAE?

%

Table will continue for vehicle group.

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm

■ Taro Pharmaceuticals U.S.A., Inc ■

L16.2.7.2 Listing of Skin Irritation Assessment

Novum Pharmaceutical Research Services Protocol / Study No. DSXS 1536 / 71515013

| Treatment Group | Patient<br>Randomization Visit<br>Number | Visit | Dermal<br>Response<br>Score | Other Effects<br>Score |
|---|---|---|---|---|
| Desoximetasone 0.25% Shampoo | xxxx-xx | Visit 1 | | Z |
| | | Visit 2 | | Z |
| | | Visit 3/Early Termination | ш | Z |

Test Vehicle Shampoo


Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm

## Novum Pharmaceutical Research Services Protocol / Study No. DSXS 1536 / 71515013

L16.2.7.3 Listing of Ocular Signs/Symptoms Assessment

| | | ٠ | | | | |
|---|---|---|---|---|---|---|
| Treatment<br>Group | Patient<br>Randomization<br>Number | Visit | Did the patient experience any ocular discomfort? | Signs/<br>Symptoms | Did the shampoo come into contact with the patient's eye? | Overall<br>Discomfort |
| Desoximetasone 0.25% Shampoo | xxxx-xx | Visit 2 | Yes | Redness/Pain | Yes | Mild |
| | | Visit 3/Early<br>Termination | °Z | | No. | |

Test Vehicle Shampoo

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm

L16.2.7.4 Listing of Positive Pregnancy Test Results

| 7 | Patient | | |
|---|---|---|---|
| l reatment | Randomization | Visit | Results |
| Group | Number | | |
| Desoximetasone 0.25% Shampoo | XXXX-XX | Visit 3/Early Termination | Positive |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm

L16.2.7.5 Listing of Abnormal Physical Examinations

| T | Patient | | | |
|---|---|---|---|---|
| l realineint | Randomization | Visit | System | Result |
| Group | Number | | | |
| Desoximetasone 0.25% Shampoo | xxxx-xx | Visit 1 | XXXXXXX | Abnormal (xxxxx) |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71515013\PDF\xxx Created on: ddmmmyy hh:mm

### NOVUM PHARMACEUTICAL RESEARCH SERVICES STATISTICAL ANALYSIS PLAN

Desoximetasone 0.25% Shampoo

Protocol / Study No. DSXS 1536 / 71515013

### 10. APPENDICES

### Appendix A: Investigator's Global Assessment (IGA) of Disease Severity of Scalp Psoriasis

| Score | Category | Description |
|---|---|---|
| 0 | Clear | Plaque elevation: no evidence of plaque elevation above normal skin |
| | | level. |
| | | Scaling: no evidence of scaling |
| | | Erythema: no redness |
| 1 | Minimal | Plaque elevation: very slight elevation above normal skin level, easier felt |
| | | than seen |
| | | Scaling: limited amount of very fine scales partially covers some of the |
| | | plaques |
| | | Erythema: very few of the plaques are light red |
| 2 | Mild | Plaque elevation: slight but definite elevation above the normal skin level, |
| | | typically with edges that are indistinct or sloped on some of the plaques. |
| | | Scaling: mainly fine scales, some plaques are partially covered. |
| | | Erythema: some plaques are light red |
| 3 | Moderate | Plaque elevation: moderate elevation with rounded or sloped edges on |
| | | most of the plaques |
| | * | Scaling: somewhat coarser scales; most plaques are partially covered. |
| | | Erythema: most plaques are red |
| 4 | Severe | Plaque elevation: marked to very marked elevation, with hard to very |
| | | hard sharp edges on virtually all or all of the plaques. |
| | | Scaling: coarse, thick scales; virtually all or all plaques are covered; |
| | | rough surface. |
| | | Erythema: virtually all or all plaques are bright to dusky red. |

### NOVUM PHARMACEUTICAL RESEARCH SERVICES STATISTICAL ANALYSIS PLAN

### Desoximetasone 0.25% Shampoo

Protocol / Study No. DSXS 1536 / 71515013

### Appendix B: Skin Assessment (Forehead, Neck and Ears)

At each clinic visit, the Investigator will evaluate the scalp and the adjacent skin (head, neck and ears) for irritation using the following scale:

### **Dermal Response and Other Effects Scoring**

### **Dermal Response**

- 0 = no evidence of irritation
- 1 = minimal erythema, barely perceptible
- 2 = definite erythema, readily visible; minimal edema or minimal papular response
- 3 =erythema and papules
- 4 = definite edema
- 5 = erythema, edema, and papules
- 6 = vesicular eruption
- 7 = strong reaction spreading beyond the application site

### **Other Effects**

- N = No other observations (numerical score = 0)
- A = Slightly glazed appearance (numerical score = 0)
- B = Marked glazed appearance (numerical score = 1)
- C = Glazing with peeling and cracking (numerical score = 2)
- F = Glazing with fissures (numerical score = 3)
- G = Film of dried serous exudates covering all or part of the application site (numerical score = 3)
- H = Small petechial erosions and/or scabs (numerical score = 3)

### NOVUM PHARMACEUTICAL RESEARCH SERVICES STATISTICAL ANALYSIS PLAN

Desoximetasone 0.25% Shampoo

Protocol / Study No. DSXS 1536 / 71515013

### **Appendix C: Ocular Discomfort Assessment**

At Visits 2 and 3 the patient will be asked to assess if any ocular discomfort was experienced, YES or NO, since the last clinic visit.

If YES is reported, the patient will be asked to report the signs and symptoms that apply from the list below or indicate any OTHER signs and symptoms experienced:

Redness

Stinging

Itching

Blur (decrease in vision)

Pain

Increased sensitivity

Swelling

Watery eyes

Burning

Spots, flashes and floaters

Eye Discharge

Foreign body sensation

In addition, the patient will be asked to indicate if the shampoo came into contact with their eye, YES or NO, since the last clinic visit. If YES is reported, the patient will be asked to rate the discomfort at the time of contact as None, Mild, Moderate or Severe.